CLINICAL TRIAL: NCT00470184
Title: Phase II Study of Capecitabine in Combination With Oxaliplatin and Radiotherapy for Esophageal and Gastroesophageal Junction Cancer
Brief Title: Oxaliplatin, Capecitabine, and Radiation Therapy in Patients Undergoing Surgery for Stage II, III, IV Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000543376; RPCI-I-64105 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-09

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Capecitabine; Oxaliplatin; Gene Expression Profiling; Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction; Chemotherapy, Adjuvant; Biopsy; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemo (Experimental): Oxaliplatin 85 mg/m2 will be administered IV on days 1, 15 and 29. Capecitabine 1250 mg/m2 will be administered in 2 divided daily doses P0 or via enteral tube, on radiation days only (Monday- Friday/ weekly). Capecitabine will be continued until the final dose of radiotherapy
  Interventions: Drug: capecitabine; Drug: oxaliplatin; Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: reverse transcriptase-polymerase chain reaction; Procedure: adjuvant therapy; Procedure: biopsy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Procedure: quality-of-life assessment; Radiation: radiation therapy

INTERVENTIONS:
Drug: capecitabine — Oral
Drug: oxaliplatin — IV
Genetic: gene expression analysis — Correlative Study
Genetic: microarray analysis — Correlative Study
Genetic: reverse transcriptase-polymerase chain reaction — Correlative Study
Procedure: adjuvant therapy — Metastatic growth control
Procedure: biopsy — Examination of tissue type
Procedure: conventional surgery — Tissue removal
Procedure: neoadjuvant therapy — Tumor shrinkage
Procedure: quality-of-life assessment — Correlative Study
Radiation: radiation therapy — Undergoing radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving oxaliplatin and capecitabine together with radiation therapy works in treating patients undergoing surgery for stage II, stage III, or stage IV esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete pathologic response (complete response [CR]) rate in patients with stage II-IVA esophageal cancer treated with neoadjuvant oxaliplatin, capecitabine, and radiotherapy.

Secondary

* Determine the clinical efficacy and toxicity of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.
* Identify basal expression and changes in gene expression that relate to CR, relapse, and survival of patients treated with this regimen.

OUTLINE:

* Neoadjuvant chemoradiotherapy: Patients receive oxaliplatin IV over 2 hours on days 1, 15, and 29 (weeks 1, 3, and 5). Patients also undergo radiotherapy on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-38 and receive oral or enteral capecitabine twice daily on the same days they undergo radiotherapy.
* Surgery: At 4-6 weeks after completion of neoadjuvant chemoradiotherapy, patients who are eligible undergo esophagectomy.
* Adjuvant chemotherapy: Beginning 4-6 weeks after surgery, patients receive oxaliplatin IV over 2 hours on days 1, 15, and 29 and oral or enteral capecitabine twice daily on days 1-5, 8-12, 15-19, 22-26, and 29. Treatment repeats approximately every 14 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor biopsies periodically. Collected samples are analyzed by gene expression studies, microarray analysis, and real-time quantitative reverse transcriptase-PCR to identify basal expression and changes in gene expression.

Quality of life is assessed periodically.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of squamous cell carcinoma of the esophagus or adenocarcinoma of the esophagus

  * Stage II-IVA disease as determined by clinical staging, including endoscopy and CT scan with or without endoscopic ultrasound
  * Bulk of gastroesophageal junction tumor should be in the esophagus
* Bronchoscopy with biopsy and cytology required if primary esophageal cancer is < 26 cm from incisors
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 4 months
* WBC > 4,000/mm³
* ANC > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 9 g/dL
* Bilirubin normal
* Creatinine normal
* AST < 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* Able to take oral medication or undergo enteral administration of medication
* No peripheral neuropathy ≥ grade 2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 90 days after completion of study treatment
* No hypersensitivity to platinum compounds, fluoropyrimidines, or antiemetics administered in combination with protocol-directed chemotherapy
* No concurrent uncontrolled illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would preclude study compliance
* No history of second malignancy except for curatively treated carcinoma in situ of the cervix or nonmelanoma skin cancer

  * Other cured tumors allowed at discretion of the principal investigator
* No known HIV or hepatitis B or C (active and/or previously treated)

PRIOR CONCURRENT THERAPY:

* No prior therapy for esophageal cancer
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-11; Primary Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Khushalani, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- COR(Capecitabine in Combination w/Oxaliplatin and Radiotherapy: Cycle 1:
  Oxaliplatin (Oxa) 85 mg/m2 IV on days (D) 1, 15 29. Capecitabine (Cap) 1250 mg/m2 in 2 divided daily doses P0 or enteral tube on radiation days (Monday- Friday/weekly), and continued until final dose of radiotherapy. Radiation administered as 1.8 Gy in 28 fractions starting on day 1. Four to six weeks after completion of Cycle I chemoradiotherapy, eligible patients will undergo esophagectomy. Cycles 2 and 3: Postoperatively, in the absence of progression, patients will be eligible for cycles 2 and 3. Cycle 2 will commence at minimum 4 to 6 weeks post-operatively, but no later than 12 weeks post-operatively. Cycles 2 and 3 will consist of OXA and CAP in the same dosage as that last administered during cycle 1. During cycles 2 and 3, CAP will be administered on days 1-29 (Monday- Friday/ weekly) and oxaliplatin on days 1, 15, 29. A minimum of 2 weeks is recommended between cycles 2 and 3.
Period: Overall Study
Arm/Group | COR(Capecitabine in Combination w/Oxaliplatin and Radiotherapy
Started | 41
Treated With Study Therapy | 36
Completed | 19
Not Completed | 22
Not completed — Not Treated(became ineligible) | 4
Not completed — Not treated (other) | 1
Not completed — disease Progression | 4
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 4
Not completed — other | 5
Not completed — recurrence | 1

BASELINE CHARACTERISTICS:
Population: treated patients
Arm/Group | COR(Capecitabine in Combination w/Oxaliplatin and Radiotherapy
Number analyzed (Participants) | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 59.53 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Time Frame: 5.5 weeks
Population: Evaluable Patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | COR(Capecitabine in Combination w/Oxaliplatin and Radiotherapy
Number analyzed (Participants) | 36
percentage of patients | 27.78 [14.20 to 45.19]

2. Secondary Outcome: Overall Response Rate (Complete and Partial Response) as Measured by RECIST Criteria After Course 1
Time Frame: 5.5 weeks
Population: evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- COR (Capecitabine in Combination w/Oxaliplatin & Radiotherapy: Cycle 1:
  Oxaliplatin (Oxa) 85 mg/m2 IV on days (D) 1, 15 29. Capecitabine (Cap) 1250 mg/m2 in 2 divided daily doses P0 or enteral tube on radiation days (Monday- Friday/weekly), and continued until final dose of radiotherapy. Radiation administered as 1.8 Gy in 28 fractions starting on day 1. Four to six weeks after completion of Cycle I chemoradiotherapy, eligible patients will undergo esophagectomy. Cycles 2 and 3: Postoperatively, in the absence of progression, patients will be eligible for cycles 2 and 3. Cycle 2 will commence at minimum 4 to 6 weeks post-operatively, but no later than 12 weeks post-operatively. Cycles 2 and 3 will consist of OXA and CAP in the same dosage as that last administered during cycle 1. During cycles 2 and 3, CAP will be administered on days 1-29 (Monday- Friday/ weekly) and oxaliplatin on days 1, 15, 29. A minimum of 2 weeks is recommended between cycles 2 and 3.
Arm/Group | COR (Capecitabine in Combination w/Oxaliplatin & Radiotherapy
Number analyzed (Participants) | 36
percentage of patients | 58.33 [40.76 to 74.49]

3. Secondary Outcome: Median Time to Progression
Time Frame: 5.5 weeks
Population: Evaluable patients
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | COR (Capecitabine in Combination w/Oxaliplatin & Radiotherapy
Number analyzed (Participants) | 36
months | NA [25.1 to NA] — NA (not available): median PFS was not reached but is >69.9 months, as is the upper bound of the 95% CI.

4. Secondary Outcome: Quality of Life Improved Rate
Time Frame: 5.5 weeks
Population: evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | COR (Capecitabine in Combination w/Oxaliplatin & Radiotherapy
Number analyzed (Participants) | 36
percentage of patients | 66.67 [49.03 to 81.44]

ADVERSE EVENTS:
Arm/Group | COR(Capecitabine in Combination w/Oxaliplatin and Radiotherapy
Serious Adverse Events (participants affected / at risk) | 12/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COR(Capecitabine in Combination w/Oxaliplatin and Radiotherapy (N=36)
Pericardial effusion - Grade 3 (Cardiac disorders) | 1 (1)
Pericarditis - Grade 2 (Cardiac disorders) | 1 (1)
Intestinal obstruction - Grade 3 (Gastrointestinal disorders) | 1 (1)
Oesophageal fistula - Grade 3 (Gastrointestinal disorders) | 1 (1)
Oesophagitis - Grade 3 (Gastrointestinal disorders) | 2 (2)
Small intestinal stenosis - Grade 3 (Gastrointestinal disorders) | 1 (1)
Death - Grade 5 (General disorders) | 1 (1)
Fatigue - Grade 3 (General disorders) | 1 (1)
Infection - Grade 3 (Infections and infestations) | 1 (1)
Pneumonia - Grade 3 (Infections and infestations) | 1 (1)
Wound infection - Grade 3 (Infections and infestations) | 1 (1)
Anastomotic leak - Grade 3 (Injury, poisoning and procedural complications) | 2 (2)
Platelet count decreased - Grade 2 (Investigations) | 1 (1)
Flank pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastasis - Grade 4 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aspiration - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COR(Capecitabine in Combination w/Oxaliplatin and Radiotherapy (N=36)
Anaemia - Grade 1 (Blood and lymphatic system disorders) | 9 (12)
Anaemia - Grade 2 (Blood and lymphatic system disorders) | 3 (3)
Anaemia - Grade 4 (Blood and lymphatic system disorders) | 1 (1)
Leukopenia - Grade 1 (Blood and lymphatic system disorders) | 16 (43)
Leukopenia - Grade 2 (Blood and lymphatic system disorders) | 10 (19)
Leukopenia - Grade 3 (Blood and lymphatic system disorders) | 4 (5)
Lymphopenia - Grade 1 (Blood and lymphatic system disorders) | 30 (81)
Lymphopenia - Grade 2 (Blood and lymphatic system disorders) | 33 (114)
Lymphopenia - Grade 3 (Blood and lymphatic system disorders) | 25 (51)
Lymphopenia - Grade 4 (Blood and lymphatic system disorders) | 6 (7)
Neutropenia - Grade 1 (Blood and lymphatic system disorders) | 3 (3)
Neutropenia - Grade 2 (Blood and lymphatic system disorders) | 5 (9)
Neutropenia - Grade 3 (Blood and lymphatic system disorders) | 2 (3)
Thrombocytopenia - Grade 1 (Blood and lymphatic system disorders) | 8 (10)
Arrhythmia - Grade 1 (Cardiac disorders) | 1 (1)
Atrial fibrillation - Grade 2 (Cardiac disorders) | 4 (4)
Palpitations - Grade 2 (Cardiac disorders) | 1 (1)
Sinus tachycardia - Grade 2 (Cardiac disorders) | 1 (1)
Tachycardia - Grade 1 (Cardiac disorders) | 1 (1)
Eye discharge - Grade 1 (Eye disorders) | 1 (1)
Photopsia - Grade 1 (Eye disorders) | 1 (1)
Vision blurred - Grade 1 (Eye disorders) | 3 (3)
Visual disturbance - Grade 1 (Eye disorders) | 1 (1)
Abdominal distension - Grade 2 (Gastrointestinal disorders) | 2 (2)
Abdominal pain - Grade 1 (Gastrointestinal disorders) | 9 (10)
Abdominal pain - Grade 2 (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper - Grade 1 (Gastrointestinal disorders) | 5 (5)
Abdominal pain upper - Grade 2 (Gastrointestinal disorders) | 1 (1)
Ascites - Grade 2 (Gastrointestinal disorders) | 1 (2)
Constipation - Grade 1 (Gastrointestinal disorders) | 16 (24)
Constipation - Grade 2 (Gastrointestinal disorders) | 2 (2)
Diarrhoea - Grade 1 (Gastrointestinal disorders) | 23 (54)
Diarrhoea - Grade 2 (Gastrointestinal disorders) | 6 (9)
Dry mouth - Grade 1 (Gastrointestinal disorders) | 1 (1)
Dyspepsia - Grade 1 (Gastrointestinal disorders) | 5 (7)
Dyspepsia - Grade 2 (Gastrointestinal disorders) | 3 (3)
Dysphagia - Grade 1 (Gastrointestinal disorders) | 8 (9)
Dysphagia - Grade 2 (Gastrointestinal disorders) | 5 (6)
Dysphagia - Grade 3 (Gastrointestinal disorders) | 2 (2)
Eructation - Grade 1 (Gastrointestinal disorders) | 2 (3)
Flatulence - Grade 1 (Gastrointestinal disorders) | 3 (3)
Flatulence - Grade 2 (Gastrointestinal disorders) | 1 (1)
Gastritis - Grade 1 (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage - Grade 2 (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying - Grade 1 (Gastrointestinal disorders) | 1 (1)
Mouth ulceration - Grade 1 (Gastrointestinal disorders) | 1 (1)
Nausea - Grade 1 (Gastrointestinal disorders) | 23 (52)
Nausea - Grade 2 (Gastrointestinal disorders) | 8 (11)
Odynophagia - Grade 1 (Gastrointestinal disorders) | 3 (3)
Oesophageal pain - Grade 1 (Gastrointestinal disorders) | 2 (2)
Oesophageal stenosis - Grade 2 (Gastrointestinal disorders) | 1 (1)
Oesophageal stenosis - Grade 3 (Gastrointestinal disorders) | 1 (1)
Oesophagitis - Grade 1 (Gastrointestinal disorders) | 5 (5)
Oesophagitis - Grade 2 (Gastrointestinal disorders) | 7 (8)
Pancreatic insufficiency - Grade 3 (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage - Grade 1 (Gastrointestinal disorders) | 1 (1)
Reflux oesophagitis - Grade 1 (Gastrointestinal disorders) | 1 (1)
Stomatitis - Grade 1 (Gastrointestinal disorders) | 1 (1)
Vomiting - Grade 1 (Gastrointestinal disorders) | 19 (31)
Vomiting - Grade 2 (Gastrointestinal disorders) | 7 (9)
Asthenia - Grade 1 (General disorders) | 1 (1)
Asthenia - Grade 2 (General disorders) | 1 (1)
Chest discomfort - Grade 1 (General disorders) | 1 (1)
Chest pain - Grade 1 (General disorders) | 2 (2)
Chest pain - Grade 2 (General disorders) | 2 (2)
Chills - Grade 1 (General disorders) | 7 (7)
Early satiety - Grade 2 (General disorders) | 1 (1)
Fatigue - Grade 1 (General disorders) | 27 (49)
Fatigue - Grade 2 (General disorders) | 12 (16)
Fibrosis - Grade 2 (General disorders) | 1 (1)
Infusion site reaction - Grade 1 (General disorders) | 1 (1)
Injection site pain - Grade 1 (General disorders) | 1 (2)
Injection site phlebitis - Grade 1 (General disorders) | 1 (1)
Injection site phlebitis - Grade 2 (General disorders) | 1 (1)
Injection site reaction - Grade 1 (General disorders) | 7 (8)
Injection site reaction - Grade 2 (General disorders) | 1 (2)
Malaise - Grade 2 (General disorders) | 1 (1)
Mucosal inflammation - Grade 1 (General disorders) | 4 (4)
Oedema peripheral - Grade 1 (General disorders) | 2 (3)
Pain - Grade 1 (General disorders) | 3 (3)
Pyrexia - Grade 1 (General disorders) | 6 (6)
Pyrexia - Grade 2 (General disorders) | 3 (3)
Systemic inflammatory response syndrome - Grade 3 (General disorders) | 1 (1)
Hyperbilirubinaemia - Grade 1 (Hepatobiliary disorders) | 1 (2)
Hyperbilirubinaemia - Grade 2 (Hepatobiliary disorders) | 3 (5)
Hyperbilirubinaemia - Grade 3 (Hepatobiliary disorders) | 4 (4)
Hypersensitivity - Grade 3 (Immune system disorders) | 2 (2)
Bronchitis - Grade 2 (Infections and infestations) | 1 (1)
Candidiasis - Grade 1 (Infections and infestations) | 1 (1)
Eye infection - Grade 1 (Infections and infestations) | 1 (1)
Fungal infection - Grade 2 (Infections and infestations) | 1 (1)
Gastroenteritis - Grade 2 (Infections and infestations) | 1 (1)
Infection - Grade 1 (Infections and infestations) | 1 (1)
Infection - Grade 2 (Infections and infestations) | 3 (3)
Infection - Grade 3 (Infections and infestations) | 4 (5)
Opportunistic infection - Grade 3 (Infections and infestations) | 1 (1)
Pneumonia - Grade 3 (Infections and infestations) | 1 (1)
Upper respiratory tract infection - Grade 1 (Infections and infestations) | 1 (1)
Anastomotic leak - Grade 1 (Injury, poisoning and procedural complications) | 2 (2)
Incision site complication - Grade 3 (Injury, poisoning and procedural complications) | 1 (1)
Seroma - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase - Grade 1 (Investigations) | 4 (4)
Alanine aminotransferase - Grade 2 (Investigations) | 3 (3)
Alanine aminotransferase decreased - Grade 1 (Investigations) | 1 (1)
Alanine aminotransferase increased - Grade 1 (Investigations) | 13 (18)
Alanine aminotransferase increased - Grade 2 (Investigations) | 9 (12)
Alanine aminotransferase increased - Grade 3 (Investigations) | 1 (1)
Aspartate aminotransferase - Grade 1 (Investigations) | 7 (16)
Aspartate aminotransferase - Grade 2 (Investigations) | 4 (5)
Aspartate aminotransferase - Grade 3 (Investigations) | 1 (1)
Aspartate aminotransferase decreased - Grade 1 (Investigations) | 1 (1)
Aspartate aminotransferase increased - Grade 1 (Investigations) | 28 (51)
Aspartate aminotransferase increased - Grade 2 (Investigations) | 13 (18)
Aspartate aminotransferase increased - Grade 3 (Investigations) | 6 (7)
Blood albumin decreased - Grade 1 (Investigations) | 4 (6)
Blood albumin decreased - Grade 2 (Investigations) | 7 (8)
Blood albumin decreased - Grade 3 (Investigations) | 4 (5)
Blood alkaline phosphatase - Grade 1 (Investigations) | 14 (27)
Blood alkaline phosphatase - Grade 2 (Investigations) | 4 (4)
Blood alkaline phosphatase increased - Grade 1 (Investigations) | 9 (9)
Blood alkaline phosphatase increased - Grade 2 (Investigations) | 2 (2)
Blood alkaline phosphatase increased - Grade 3 (Investigations) | 1 (1)
Blood bilirubin - Grade 1 (Investigations) | 4 (4)
Blood bilirubin - Grade 2 (Investigations) | 1 (1)
Blood calcium decreased - Grade 1 (Investigations) | 2 (2)
Blood calcium decreased - Grade 2 (Investigations) | 5 (5)
Blood calcium increased - Grade 1 (Investigations) | 1 (1)
Blood creatine increased - Grade 1 (Investigations) | 1 (1)
Blood creatine phosphokinase - Grade 1 (Investigations) | 1 (1)
Blood creatinine - Grade 1 (Investigations) | 5 (6)
Blood creatinine - Grade 2 (Investigations) | 1 (1)
Blood glucose decreased - Grade 1 (Investigations) | 2 (2)
Blood glucose increased - Grade 1 (Investigations) | 6 (6)
Blood glucose increased - Grade 2 (Investigations) | 2 (2)
Blood glucose increased - Grade 3 (Investigations) | 1 (1)
Blood potassium decreased - Grade 1 (Investigations) | 4 (4)
Blood potassium increased - Grade 1 (Investigations) | 2 (3)
Blood potassium increased - Grade 2 (Investigations) | 2 (2)
Blood sodium decreased - Grade 1 (Investigations) | 7 (8)
Blood sodium increased - Grade 1 (Investigations) | 3 (3)
Haemoglobin - Grade 1 (Investigations) | 26 (57)
Haemoglobin - Grade 2 (Investigations) | 12 (32)
Haemoglobin - Grade 3 (Investigations) | 2 (2)
Haemoglobin decreased - Grade 1 (Investigations) | 7 (8)
Haemoglobin decreased - Grade 2 (Investigations) | 4 (4)
Lymphocyte count decreased - Grade 1 (Investigations) | 1 (1)
Lymphocyte count decreased - Grade 2 (Investigations) | 2 (2)
Platelet count - Grade 1 (Investigations) | 1 (1)
Platelet count decreased - Grade 1 (Investigations) | 26 (52)
Platelet count decreased - Grade 2 (Investigations) | 5 (8)
Transaminases increased - Grade 2 (Investigations) | 1 (1)
Troponin I - Grade 3 (Investigations) | 1 (1)
Weight decreased - Grade 1 (Investigations) | 7 (8)
Weight decreased - Grade 2 (Investigations) | 12 (13)
Weight decreased - Grade 3 (Investigations) | 3 (4)
White blood cell count decreased - Grade 1 (Investigations) | 7 (9)
White blood cell count decreased - Grade 2 (Investigations) | 3 (3)
Anorexia - Grade 1 (Metabolism and nutrition disorders) | 13 (18)
Anorexia - Grade 2 (Metabolism and nutrition disorders) | 10 (14)
Anorexia - Grade 3 (Metabolism and nutrition disorders) | 3 (3)
Dehydration - Grade 2 (Metabolism and nutrition disorders) | 6 (6)
Gout - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia - Grade 1 (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia - Grade 1 (Metabolism and nutrition disorders) | 19 (34)
Hyperglycaemia - Grade 2 (Metabolism and nutrition disorders) | 11 (18)
Hyperglycaemia - Grade 3 (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia - Grade 1 (Metabolism and nutrition disorders) | 6 (7)
Hypermagnesaemia - Grade 1 (Metabolism and nutrition disorders) | 10 (24)
Hypermagnesaemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesaemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia - Grade 1 (Metabolism and nutrition disorders) | 8 (13)
Hypernatraemia - Grade 2 (Metabolism and nutrition disorders) | 2 (3)
Hypernatraemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia - Grade 1 (Metabolism and nutrition disorders) | 13 (29)
Hypoalbuminaemia - Grade 2 (Metabolism and nutrition disorders) | 21 (33)
Hypoalbuminaemia - Grade 3 (Metabolism and nutrition disorders) | 3 (6)
Hypocalcaemia - Grade 1 (Metabolism and nutrition disorders) | 11 (19)
Hypocalcaemia - Grade 2 (Metabolism and nutrition disorders) | 9 (10)
Hypocalcaemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia - Grade 1 (Metabolism and nutrition disorders) | 6 (6)
Hypoglycaemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia - Grade 1 (Metabolism and nutrition disorders) | 9 (15)
Hypokalaemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia - Grade 3 (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia - Grade 1 (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesaemia - Grade 2 (Metabolism and nutrition disorders) | 6 (6)
Hyponatraemia - Grade 1 (Metabolism and nutrition disorders) | 20 (56)
Hyponatraemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia - Grade 1 (Metabolism and nutrition disorders) | 3 (3)
Hypophosphataemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Back pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 5 (6)
Back pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 3 (3)
Gouty arthritis - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (3)
Gouty arthritis - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscular weakness - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness - Grade 1 (Nervous system disorders) | 11 (19)
Dysaesthesia - Grade 1 (Nervous system disorders) | 2 (2)
Dysgeusia - Grade 1 (Nervous system disorders) | 7 (13)
Dysgeusia - Grade 2 (Nervous system disorders) | 3 (3)
Headache - Grade 1 (Nervous system disorders) | 5 (5)
Hyperaesthesia - Grade 1 (Nervous system disorders) | 3 (3)
Hypoaesthesia - Grade 1 (Nervous system disorders) | 5 (5)
Neuroleptic malignant syndrome - Grade 3 (Nervous system disorders) | 1 (1)
Neuropathy - Grade 2 (Nervous system disorders) | 1 (1)
Paraesthesia - Grade 1 (Nervous system disorders) | 6 (6)
Paraesthesia - Grade 2 (Nervous system disorders) | 2 (2)
Paraesthesia - Grade 3 (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy - Grade 1 (Nervous system disorders) | 23 (64)
Peripheral sensory neuropathy - Grade 2 (Nervous system disorders) | 2 (2)
Peroneal nerve palsy - Grade 1 (Nervous system disorders) | 1 (1)
Restless legs syndrome - Grade 1 (Nervous system disorders) | 2 (2)
Tremor - Grade 1 (Nervous system disorders) | 1 (1)
Vocal cord paralysis - Grade 1 (Nervous system disorders) | 1 (1)
Anxiety - Grade 1 (Psychiatric disorders) | 1 (1)
Anxiety disorder - Grade 2 (Psychiatric disorders) | 1 (1)
Confusional state - Grade 2 (Psychiatric disorders) | 1 (1)
Depression - Grade 2 (Psychiatric disorders) | 2 (2)
Drug dependence - Grade 2 (Psychiatric disorders) | 1 (1)
Insomnia - Grade 1 (Psychiatric disorders) | 9 (10)
Insomnia - Grade 2 (Psychiatric disorders) | 1 (1)
Chromaturia - Grade 1 (Renal and urinary disorders) | 1 (1)
Dysuria - Grade 1 (Renal and urinary disorders) | 1 (1)
Renal failure acute - Grade 1 (Renal and urinary disorders) | 1 (1)
Aspiration - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Choking sensation - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chylothorax - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 18 (23)
Cough - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dysphonia - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Dysphonia - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 12 (15)
Dyspnoea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea exertional - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccups - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Drug eruption - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis - Grade 1 (Skin and subcutaneous tissue disorders) | 6 (7)
Hyperhidrosis - Grade 2 (Skin and subcutaneous tissue disorders) | 3 (3)
Photosensitivity reaction - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus - Grade 1 (Skin and subcutaneous tissue disorders) | 4 (7)
Pruritus - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - Grade 1 (Skin and subcutaneous tissue disorders) | 8 (10)
Rash - Grade 2 (Skin and subcutaneous tissue disorders) | 3 (3)
Rash - Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash generalised - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (2)
Skin lesion - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin odour abnormal - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis - Grade 3 (Vascular disorders) | 3 (3)
Flushing - Grade 1 (Vascular disorders) | 1 (1)
Hypertension - Grade 1 (Vascular disorders) | 1 (1)
Hypertension - Grade 3 (Vascular disorders) | 1 (1)
Hypotension - Grade 2 (Vascular disorders) | 2 (2)
Lymphorrhoea - Grade 2 (Vascular disorders) | 1 (1)
Orthostatic hypotension - Grade 1 (Vascular disorders) | 1 (1)
Orthostatic hypotension - Grade 2 (Vascular disorders) | 1 (1)
Phlebitis - Grade 2 (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes